CLINICAL TRIAL: NCT03146585
Title: Alterations of Glycocalyx in Critical Illness and During Major Surgery and Approaches for Glycocalyx Protection
Brief Title: Glycocalyx Damage in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Vladimir Cerny, Clinical Professor, University Hospital Hradec Kralove
Other Study IDs: AZVCR 9307_3
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Critical Illness
Keywords: Glycocalyx
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients on artificial ventilation
  Interventions: Device: PBR assessment
- Patients on renal replacement therapy
  Interventions: Device: PBR assessment
- Patients with targeted temperature management
  Interventions: Device: PBR assessment

INTERVENTIONS:
Device: PBR assessment — Sublingual microcirculation will be investigated by specialized handheld videomicroscopy device for PBR index.

SUMMARY:
The hypothesis to be tested: GCX damage and its dynamics correlate to various patient related factors and to using organ-supporting measures. There is a correlation between length of organ support and GCX damage.

The aim of the study: Evaluation of the relationship between GCX damage and duration of various organ supporting measures.

Type of the study: Observational. Subjects: Adult patients admitted to ICU and requiring organ supporting therapy.

Sample size: We plan enrollment of 75 patients on invasive ventilatory support in the duration of least 5 days, 50 patients on renal supporting therapy lasting at least 5 days and 20 patients with target temperature management for neuroprotection.

Intervention: none Data to be recorded and analysed: Demographics, type of patients (trauma, post surgical, medical, after cardiac arrest), severity score - Apache II, SOFA, fluid balance, presence of delirium, clinical outcome, sublingual microcirculation by SDF imaging at time points: before or at the start of organ support, after 24 hours (day 1), day 3, 5, 7 and/or at discharge or before death, microcirculatory data, and Perfused Boundary Region.

ELIGIBILITY:
Inclusion Criteria:

* adult patients admitted to ICU
* artifitial ventilation
* renal replacement therapy
* targeted temperatura management

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to ICU meeting inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Cerny, MD, PhD, FCCM, Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Třebeš, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients admitted to our ICU with any kind of organ support.
Period: Overall Study
Arm/Group | Patients on Artificial Ventilation | Patients on Renal Replacement Therapy | Patients With Targeted Temperature Management
Started | 25 | 10 | 5
Completed | 25 | 10 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients on Artificial Ventilation | Patients on Renal Replacement Therapy | Patients With Targeted Temperature Management | Total
Number analyzed (Participants) | 25 | 10 | 5 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 10 | 5 | 40
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (5) | 50 (6) | 62 (3) | 60 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 2 | 15
  Male | 15 | 7 | 3 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Czechia | 25 | 10 | 5 | 40
PBR value [Mean (Inter-Quartile Range); unit: micrometer] — The Perfused Boundary Region (PBR) is an indirect assessment of the thickness of the endothelial glycocalyx in sublingual microcirculation.
  micrometer | 2.02 [1.92 to 2.20] | 2.13 [2.02 to 2.28] | 2.07 [1.92 to 2.32] | 2.10 [2.00 to 2.20]

OUTCOME MEASURES:

1. Primary Outcome: Perfused Boundary Region (PBR) in One Week
Description: PBR is an indirect measure of assessment of the endothelial glycocalyx thickness in sublingual microcirculation.
Time Frame: One week on ICU
Measure: Median (Inter-Quartile Range); unit: micrometer
Arm/Group | Patients on Artificial Ventilation | Patients on Renal Replacement Therapy | Patients With Targeted Temperature Management
Number analyzed (Participants) | 25 | 10 | 5
micrometer | 1.95 [1.77 to 2.12] | 1.97 [1.75 to 2.12] | 2.02 [1.71 to 2.15]

ADVERSE EVENTS:
Description: Adverse events were not collected since the study is observational. If the patient died it was due to the natural course of the disease.
Arm/Group | Patients on Artificial Ventilation | Patients on Renal Replacement Therapy | Patients With Targeted Temperature Management
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT03146585/Prot_SAP_000.pdf